CLINICAL TRIAL: NCT03794570
Title: Blood Flow Restriction Therapy to Prevent Muscle Atrophy Following Anterior Cruciate Ligament Reconstruction
Brief Title: BFR Therapy After ACL Reconstruction
Acronym: BFR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator separated from institution
Sponsor: Steadman Philippon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-35
Record Dates: First submitted 2018-12-20; First posted 2019-01-07 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: ACL Injury; Quadriceps Muscle Atrophy
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Double blinded randomized control trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients and outcomes assessors will be blinded to treatment group. Physical therapy providers will not be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (Sham Comparator): Patients in this group will have BFR tourniquet applied but inflated to only minimal pressure.
  Interventions: Device: Sham blood flow restriction therapy - with Delfi Personalized Tourniquet System
- Blood Flow Restriction (BFR) Therapy (Experimental): Patients in this group will have BFR tourniquet applied and inflated to 80% limb occlusion pressure
  Interventions: Device: Blood flow restriction therapy - with Delfi Personalized Tourniquet System

INTERVENTIONS:
Device: Blood flow restriction therapy - with Delfi Personalized Tourniquet System — Physical therapy performed with Blood flow restriction therapy tourniquet inflated to 80% limb occlusion pressure
  Arms: Blood Flow Restriction (BFR) Therapy
Device: Sham blood flow restriction therapy - with Delfi Personalized Tourniquet System — Physical therapy performed with Blood flow restriction therapy tourniquet inflated to only minimal pressure
  Arms: Control

SUMMARY:
This study is a prospective, double-blinded, randomized control trial examining the effect of blood flow restriction (BFR) therapy on reducing post-operative quadriceps atrophy in patients undergoing anterior cruciate ligament reconstruction (ACLR). Following ACLR, patients will undergo a rehabilitation protocol either w/ BFR therapy or sham BFR therapy.

DETAILED DESCRIPTION:
Patients will be randomized to either BFR therapy or no BFR therapy. Randomization will be carried out using block randomization with blocks of 6.

Those undergoing BFR therapy will have a Delfi Personalized Tourniquet System (PTS) cuff applied to the proximal thigh of their operative leg and inflated to 80% limb occlusive pressure (LOP) calculated by the Delfi PTS device during physical therapy (PT) sessions from day 2 after surgery through day 7 after surgery. Those in the no BFR group will have the Delfi PTS cuff applied to their proximal thigh with inflation of the tourniquet to minimal pressure only. BFR therapy will be administered by health care providers who have undergone training and certification for BFR therapy with the Delfi PTS device.

Both groups will undergo the following PT regimen two times daily beginning on the day after the surgical procedure and lasting for 6 weeks post-operatively:

* Quad sets = x1 min isometric hold, 30 sec off, 3 sets
* Terminal knee extensions = 3x15, 30 sec rest or short arc quads sitting 1 x 30 + 3 x 15, 30 sec rest
* Once range of motion (ROM) allows: Bike 10 mins, low to no resistance

Each physical therapy visit will last approximately 60 minutes. During that time, there will be a total estimated time of 5-7 minutes during which the tourniquet cuff will be on the thigh, and the tourniquet will be inflated for a similar time period. The tourniquet will inflate for about 1 minute in order to find out the specific pressure for the patient's leg and then will remain inflated until exercises are completed, which should take 4-6 minutes. The cuff will then be deflated and is removed from the leg within about 30 seconds of being deflated.

Patients will have MRI performed pre-operatively and at 6 weeks post-operatively with axial cuts to 50% femoral length above joint line. Quadriceps cross-sectional area will be measured by a blinded observer using MRI. Patients will have clinical measurements including thigh girth, Lachman test, knee joint range of motion, and knee joint swelling performed pre-operatively, at post-op day 1, post-op day 14, and 6 weeks post-operatively. All clinical measurements will be performed by a blinded observer. Additionally, patient reported pain level will be obtained at the same timepoints in which clinical measurements are performed using visual analog scale.

In order to ensure there are no nerve injuries present in patients prior to undergoing application and inflation of thigh tourniquet, all patients in the study will have single shot adductor and/or sciatic nerve blocks to ensure 24 hour period without nerve block prior to initiation of BFR therapy. Patients included in the study cannot have a nerve block lasting longer than the day of surgery. To ensure no new nerve deficits are present, the patients will undergo a physical examination during morning rounding on post-operative day 1 to assess for new nerve deficits.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-70
* Undergoing ACL reconstruction with patellar tendon autograft
* Full weightbearing after surgery
* Surgery performed within 14 days of ACL injury
* No nerve catheter in place

Exclusion Criteria:

* Meniscal root tears
* radial meniscal tears
* multi-ligament knee injury
* revision ACL reconstruction
* concomitant osteotomies
* concomitant cartilage resurfacing procedures
* fracture preventing full-weightbearing of operated extremity
* previous history of deep vein thrombosis (DVT)
* new nerve injury/findings affecting operative extremity
* active femoral nerve catheter
* nerve block lasting longer than day of surgery
* patients unable to tolerate BFR treatment
* untolerable post-operative pain due to absence of nerve catheter
* proximal thigh girth greater than 34cm
* time to surgery greater than 14 days

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Quadriceps Cross-Sectional Area | Pre-op and 6-weeks post-operative
  Change in quadriceps cross-sectional area measured on MRI pre-operatively compared to post-operatively

SECONDARY OUTCOMES:
Numeric rating scale pain | Days 1, 14, and 6 weeks after surgery
  Patient reported pain levels using numeric rating scale (NRS) on a scale of 1-10 where 10 represents maximal pain and 1 represents minimal pain
Thigh girth | Days 1, 14, and 6 weeks after surgery
  Measured thigh girth 15cm above knee joint line
Knee joint range of motion | Days 1, 14, and 6 weeks after surgery
  Measure knee range of motion

CONTACTS AND LOCATIONS:
Locations (1):
- The Steadman Clinic, Vail, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No sharing